CLINICAL TRIAL: NCT04066231
Title: ANTERO-4: A Clinical Investigation of the Effects of Erythromycin on Gastric Motility, Assessed With the VIPUN Gastric Monitoring System in Healthy Adults
Brief Title: ANTERO-4: VIPUN Gastric Monitoring System in an Erythromycin Model
Acronym: ANTERO-4
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigational medical device no longer available
Sponsor: Prof Dr Jan Tack (Other)
Responsible Party: Sponsor-Investigator, Prof Dr Jan Tack, Head of Clinic - Gastroenterology / Professor of Medicine / Principal Investigator, Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S62862
Record Dates: First submitted 2019-08-06; First posted 2019-08-26 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Gastric Motility
MeSH Terms: interventions — erythromycin lactobionate

STUDY DESIGN:
Intervention Model Description: A gastroprokinetic agent is administered to stimulate gastric motility.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VIPUN GMS (Experimental): Single arm study.
  Interventions: Device: VIPUN GMS; Drug: Erythromycin Lactobionate

INTERVENTIONS:
Device: VIPUN GMS — Motility is measured for 4 hours with the VIPUN Gastric Monitoring System (GMS).
Drug: Erythromycin Lactobionate — Test model: Erythromycin has gastroprokinetic properties. The primary aim of this investigation is to validate the ability of the VIPUN GMS to discriminate between normal and pharmacologically-enhanced fasting gastric motility in healthy adults.
  Erythromycin Lactobionate infusion: 200 mg i.v. infusion over a period of 20 minutes. Note: Erythromycin is not labeled as a gastroprokinetic agent in Belgium.

SUMMARY:
It has been demonstrated that the VIPUN Gastric Monitoring System (GMS) can discriminate healthy physiological and pharmacologically-inhibited gastric motility, using a codeine-model in healthy adults (S60320 / AFMPS80M0687).

Erythromycin is a gastroprokinetic agent, known to stimulate gastric contractility. A single dose of 200 mg erythromycin has been shown to induce a prolonged period of enhanced phasic contractile activity.

The primary aim of this investigation is to validate the ability of the VIPUN GMS to discriminate between normal and pharmacologically-enhanced fasting gastric motility in healthy adults.

The performance of the VIPUN GMS can be enhanced by data-driven optimization of the VIPUN Motility Algorithm, used to quantify gastric motility.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Aged between and including 18 and 65 years
* BMI between and including 18 and 30
* Understand and able to read Dutch
* In good health on the basis of medical history
* Refrains from herbal, vitamin and other dietary supplements on the day of the visits

Exclusion Criteria:

* Dyspeptic symptoms (assessed with PAGI-SYM questionnaire)
* Using any medication that might affect gastric function or visceral sensitivity
* Known / suspected current use of illicit drugs
* Known psychiatric or neurological illness
* Any gastrointestinal surgery that could influence normal gastric function in the opinion of the investigator
* History of heart or vascular diseases like irregular heartbeats, angina or heart attack
* Nasopharyngeal surgery in the last 30 days
* Suspected basal skull fracture or severe maxillofacial trauma
* History of thermal or chemical injury to upper respiratory tract or esophagus
* Current esophageal or nasopharyngeal obstruction
* Known coagulopathy
* Known esophageal varices
* Pregnant or breastfeeding women
* Have known side-effects/allergic reactions when taking erythromycin or other macrolide antibiotics (such as azithromycin, clarithromycin)
* Kidney disease
* Liver disease
* Myasthenia gravis
* QT prolongation (QT ≥400 ms) at the screening
* Cardiac arrhythmia or heart failure
* History of C. difficile infection
* Family history of QT prolongation, sudden cardiac death or other heart problems
* Recent vaccinations with live bacterial vaccines (such as typhoid vaccine)
* Concomitant medication use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-09-07 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
GBMI baseline | t = 0 - 119 minutes
  Gastric Balloon Motility Index (GBMI) is measured with the VIPUN Gastric Monitoring System. GBMI is a value between 0 and 1.
GBMI120 - 139 | t = 120 - 139 minutes
  Motility during erythromycin administration. Gastric Balloon Motility Index (GBMI) is measured with the VIPUN Gastric Monitoring System. GBMI is a value between 0 and 1.

SECONDARY OUTCOMES:
GBMI140-240 | t = 140 - 240 minutes
  Motility in the period 140 - 240 minutes. Gastric Balloon Motility Index (GBMI) is measured with the VIPUN Gastric Monitoring System. GBMI is a value between 0 and 1.
Symptoms | t = 0 - 240 minutes
  Epigastric symptoms (nausea, bloating, pain) are surveyed with Visual Analogue Scales for severity of each individual symptom (100 mm, 0 = Absent to 100 mm = worst possible sensation) at a 15 minute interval.
Incidence of adverse events | t = 0 - 240 minutes
  Incidence of adverse events
Severity of adverse (device) events/effects | t = 0 - 240 minutes
  Severity of adverse (device) events/effects
Seriousness of adverse (device) events/effects | t = 0 - 240 minutes
  Seriousness of adverse (device) events/effects
Relatedness of adverse (device) events/effects | t = 0 - 240 minutes
  Relatedness of adverse (device) events/effects
Incidence of device deficiencies of the investigational medical device | t = 0 - 240 minutes
  Qualitative description of the event, onset, duration, origin, action taken and outcome of the event
Incidence of protocol deviations related to the investigational medical device | t = 0 - 240 minutes
  Qualitative description of the event, onset, duration, origin, action taken and outcome of the event

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goelen N, Tack J, Janssen P. Erythromycin stimulates phasic gastric contractility as assessed with an isovolumetric intragastric balloon pressure measurement. Neurogastroenterol Motil. 2021 Feb;33(2):e13991. doi: 10.1111/nmo.13991. Epub 2020 Oct 6. PMID 33025716